CLINICAL TRIAL: NCT04525014
Title: A Phase 1 Trial of RRx-001 in Combination With Irinotecan and Temozolomide for Pediatric Patients With Recurrent or Progressive Malignant Solid and Central Nervous System Tumors
Brief Title: RRx-001 Given With Irinotecan and Temozolomide for Pediatric Patients With Recurrent or Progressive Malignant Solid and Central Nervous System Tumors
Acronym: PIRATE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: EpicentRx, Inc. (Industry)
Collaborators: Texas Children's Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-45787
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Brain Tumor, Recurrent; Brain Tumor, Pediatric; Central Nervous System Neoplasms; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: Brain cancer; Pediatric cancer; Spinal cord tumor; Solid tumor
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Neoplasms; Spinal Cord Neoplasms | interventions — RRx-001; Temozolomide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RRx-001, Temozolomide and Irinotecan (Experimental)
  Interventions: Drug: RRx-001; Drug: Temozolomide; Drug: Irinotecan

INTERVENTIONS:
Drug: RRx-001 — RRx-001 will be administered every 3 weeks via intravenous infusion at three dose levels: 0.5 mg/m2 (Max 1 mg), 1 mg/m2 (Max 2 mg), and 2 mg/m2 (Max 4 mg).
Drug: Temozolomide — 100 mg/m2 (children ≥0.5 m2) or 3 mg/kg (children <0.5 m2) daily for 5 days beginning on day 1 of each cycle
Drug: Irinotecan — 90 mg/m2 taken orally daily for 5 days administered 1 hour after temozolomide

SUMMARY:
The PIRATE study tests the experimental drug RRx-001 in combination with 2 chemotherapy drugs that are commonly used in patients with cancer. RRx-001 has been used alone and with other anti-cancer medicines in adults. However, the investigators do not know what effects it will have in children and young adults.

DETAILED DESCRIPTION:
The goals of the PIRATE study are:

* Determine if the adult dose of RRx-001 is safe when given together with 2 chemotherapy drugs called irinotecan and temozolomide in children and young adults with previously-treated cancerous tumors
* Determine the side effects of RRx-001 in children and young adults when given together with irinotecan and temozolomide
* Understand if the combination of RRx-001, irinotecan, and temozolomide is helpful for children and young adults with previously-treated cancerous tumors
* In patients with brain tumors, measure if RRx-001 causes changes in the tumor on Magnetic Resonance Imaging (MRI)
* Determine if RRx-001 causes changes in the immune system which may help the body naturally fight the tumor

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent or progressive malignant (World Health Organization (WHO) grade 3 or 4 tumors) primary brain or spinal cord tumors and solid tumors (excluding lymphomas)
2. Eligible patients may have measureable or non-measurable but evaluable disease according to the reviewed Response Evaluation Criteria in Solid Tumors (RECIST) guidelines version 1.1 criteria.
3. Patients must have a Karnofsky score of ≥50% if >16 years old or a Lansky score of ≥50 if ≤16 years old
4. Patients must have fully recovered from the acute treatment-related toxicities (defined as <grade 1) of their most recent prior anti-neoplastic therapy prior to study enrollment.
5. Patients must be at least 4 weeks from major surgery including craniotomy or tumor debulking/resection and at least 1 week from stereotactic biopsy prior to study enrollment. Patients must have fully recovered from all acute effects of prior surgical intervention excluding central line placement prior to study enrollment. Patients must have fully recovered from all acute effects of central line placement prior to initiation of study treatment.
6. Patients with neurological deficits should have deficits that are stable for a minimum of 7 days prior to study enrollment. Patients with seizure disorders may be enrolled if the seizures are well-controlled with a stable seizure frequency and duration for a minimum 7 days.
7. Patients on chronic systemic steroids must be on a stable or decreasing dose for at least 7 days prior to study enrollment. If used to modify immune adverse events related to prior therapy, ≥ 14 days must have elapsed since last dose of corticosteroid.
8. Platelet count ≥75,000/mm3. Patient must be transfusion independent defined as not receiving platelet transfusions with a 7-day period prior to study enrollment.
9. Peripheral absolute neutrophil count ≥1000/mm3
10. Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2 or a serum creatinine based on age and sex
11. Conjugated bilirubin ≤1.5 times the institutional laboratory's upper limit of normal
12. Alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase (SGPT)) ≤3 times the institutional laboratory's upper limit of normal
13. Aspartate transaminase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) ≤3 times the institutional laboratory's upper limit of normal
14. Adequate pulmonary function defined as:
15. Oxygen saturation as measured by pulse oximetry > 93% on room air
16. No evidence of dyspnea at rest
17. Left ventricular ejection fraction > 50%
18. Patients of child-bearing potential of both genders must utilize contraception including but not limited to hormonal contraception, barrier method, or abstinence for the duration of the study and 28 days after completion of study.
19. Patients must have a central line in place prior to administration of the first dose of RRx-001. Patients must have fully recovered from all acute effects of central line placement prior to initiation of study treatment.
20. The patient or parent/legally authorized representative is able to understand the consent and is willing to sign a written informed consent document according to institutional guidelines. Assent, when appropriate, will be obtained according to institutional guidelines.
21. Patients must be able to safely take oral medications either as liquid or tablet.

Exclusion Criteria:

1. Pregnant or breast feeding females
2. Patients with the following conditions will be excluded from study enrollment: cyanotic heart disease, intermediate or severe β-thalassemia, known glucose-6-phosphate dehydrogenase (G6PD) deficiency, active infections, concurrent malignancy, a known thrombophilia syndrome, or a personal history of venous thromboembolism including catheter-associated thrombi.31-34 Additionally, patients with clinically significant or poorly controlled cardiac, pulmonary, hepatic, or other organ dysfunction that, in the opinion of the investigator, would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity, or interfere with the study procedures or results are not eligible for study enrollment. Patients with a known coagulopathy or bleeding diathesis or who have undergone either a solid organ or allogeneic bone marrow/stem cell transplant are not eligible for study enrollment.
3. Patients taking concurrent anti-cancer or investigational drug therapies are not eligible for study enrollment.
4. Patients taking anti-oxidants including alpha lipoic acid, vitamin E, N- acetylcysteine, and omega 3 fatty acid supplements are not eligible for study enrollment. Patients must be off these drugs for a minimum of 7 days prior to study enrollment and must remain off anti-oxidant medications for the duration of study treatment.
5. While on study, concomitant use of clozapine, echinacea, leflunomide, natalizumab, and tofacitinib are prohibited due to potential for increased temozolomide toxicity.
6. Patients who have received drugs that are strong inducers of CYP3A4 within 14 days prior to study enrollment are not eligible.
7. Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to drug administration plan, other study procedures, and study restrictions are not eligible for study enrollment.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose | 18 months
  Estimate the recommended phase 2 dose of RRx-001 administered every 3 weeks as an IV infusion in combination with oral irinotecan and temozolomide in pediatric patients with recurrent or progressive malignant solid or central nervous system (CNS) tumors.

OTHER OUTCOMES:
Grade 3 or higher CTCAE version 5.0 adverse event terms | 18 months
  Describe the toxicities of RRx-001 in combination with irinotecan and temozolomide administered on this schedule in this population.
Progression-free survival (PFS) | 15 months
  Describe the anti-tumor effects of RRx-001 in combination with irinotecan and temozolomide administered on this schedule in this population in the context of a Phase 1 trial.
Overall survival (OS) | 15 months
  Describe the anti-tumor effects of RRx-001 in combination with irinotecan and temozolomide administered on this schedule in this population in the context of a Phase 1 trial.
Summarize tumor response rates | 15 months
  Imaging-based evaluation is preferred to evaluation by clinical examination unless the lesion(s) being followed cannot be imaged but are assessable by clinical exam.
Change in tumor perfusion | 15 months
  Measure treatment-induced change in tumor perfusion
Response correlation for change in tumor perfusion | 15 months
  Correlation of change in tumor perfusion to matched patient's best treatment response
Change in cellularity | 15 months
  Measure treatment-induced change in cellularity
Response correlation for change in cellularity | 15 months
  Correlation of change in cellularity to matched patient's best treatment response
Ratio of M1 to M2 peripheral blood circulating monocytes | 5 months
  Assess for change in the ratio of M1 to M2 peripheral blood circulating monocytes over the first 5 cycles of therapy.
Response correlation for ratio of M1 to M2 peripheral blood circulating monocytes | 5 months
  Correlation of change in the ratio of M1 to M2 peripheral blood circulating monocytes over the first 5 cycles of therapy to matched patient's best treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Oronsky, MD, Study Director — EpicentRx, Inc.; Stephanie Fetzko, MD, Principal Investigator — Texas Children's Cancer Center
Locations (1):
- Texas Children's Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No